CLINICAL TRIAL: NCT04884503
Title: Assessment of the Effectiveness of the Selected Treatment Method and Psychological Disorders of Primary Burning Mouth Syndrome
Brief Title: Evaluation of the Effectiveness of the Selected Method of Treatment of Primary Burning Mouth Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kb668/2018
Record Dates: First submitted 2021-04-27; First posted 2021-05-13 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-05

CONDITIONS: Burning Mouth Syndrome; Glossodynia
Keywords: BMS, , clonazepam, BMS psychological disturbance
MeSH Terms: conditions — Burning Mouth Syndrome; Glossalgia | interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients diagnosed with BMS traeting with Clonazepam (Experimental): Dosing of clonazepam was as follows: in the first week, 1 mg to be sucked for 2 minutes, then swallowed (once a day in the morning), in the second week, 1 mg to be sucked for 2 minutes, and then swallowed (twice a day in the morning and one hour before falling asleep), in the third week, 1 mg to be sucked for 2 minutes and in the fourth week 1 mg to be sucked for 2 minutes, then swallowed (once a day in the morning)
  Interventions: Drug: Clonazepam tablets
- Patients diagnosed with BMS treating with tongue pads (Active Comparator): patients wearing tongue pads 3 times a day for 20 minutes for 4 weeks to exclude parafunctions
  Interventions: Device: tongue pads

INTERVENTIONS:
Drug: Clonazepam tablets — Dosing of clonazepam was as follows: in the first week, 1 mg to be sucked for 2 minutes, then swallowed (once a day in the morning), in the second week, 1 mg to be sucked for 2 minutes, and then swallowed (twice a day in the morning and one hour before falling asleep), in the third week, 1 mg to be sucked for 2 minutes and in the fourth week 1 mg to be sucked for 2 minutes, then swallowed (once a day in the morning)
  Other Names: patients treating with clonazepam
  Arms: Patients diagnosed with BMS traeting with Clonazepam
Device: tongue pads — wearing a tongue pad 3 times a day for 20 minutes for 4 weeks
  Other Names: patients treating with tonque pads
  Arms: Patients diagnosed with BMS treating with tongue pads

SUMMARY:
The burning mouth syndrome (BMS) is a chronic pain syndrome of the oral mucosa. Feels like experiencing a burning sensation, pain, stinging, or numbness in the mouth along with a feeling of dryness, paraesthesia, taste disturbance or hypersensitivity.The complaints are usually bilateral, of moderate intensity, they persist for a minimum of 4-6 months and concern the clinically unchanged membrane mucous.The psychiatric aspect of BMS is very important. The presence of BMS has been shown to be associated with depression, increased anxiety levels, hypochondria, and carcinophobia and emotional instability

DETAILED DESCRIPTION:
The burning mouth syndrome (BMS) is a chronic pain syndrome of the oral mucosa. Patients have experiencing a burning sensation, pain, stinging, or numbness in the mouth along with a feeling of dryness, paraesthesia, taste disturbance or hypersensitivity. The complaints are usually bilateral, of moderate intensity, they persist for a minimum of 4-6 months and concern the clinically unchanged membrane mucous.The psychiatric aspect of BMS is very important. The presence of BMS has been shown to be associated with depression, increased anxiety levels, hypochondria, and carcinophobia and emotional instability

The first step is to determine the specific type of BMS, i.e. to exclude a causal relationship with the existing local factors, general diseases and medications taken.

The pathophysiology of Primary Burning Mouth Syndrome is unclear. Due to the lack of morphological changes in the oral cavity with the simultaneous occurrence of troublesome pain symptoms, it is now assumed that pain in BMS has a neuropathic mechanism.

Among the psychotropic drugs, the most commonly used in the treatment of BMS was clonazepam, a drug with anticonvulsant and anxiolytic properties .

In this study, the investigators used clonazepam because of which it has proven effectiveness in therapy in combination with a tongue protector made for the purpose of the test. Use of a tongue protector in the form of a bag put on it 3 times a day is relatively new method of treatment, which is to exclude the detachment of the tongue's para-function on burning.

60 patients were qualified for the study, of which 57 patients, including 34 women and 23 men, aged 47-77 years, took part in the program.

Pain assessment The symptoms of pain intensity BMS were assessed using the VAS (Visual Analog Scale) The duration of burning was also assessed, the type of burning according to Levis, the occurrence of taste disturbances and their determination, subjective feeling of dry mouth, place of burning sensation: tongue, palate, lips, mucosa of the mouth vestibule with gums, cheek mucosa The psychologist cooperating in the project conducted and then interpreted four psychological tests: STAI (state and trait anxiety inventory) and the Beck Anxiety Scale BAI and the Beck Depression Scale BDI. Moreover, the WHOQOL quality of life test was carried out - according to WHO

A follow-up examination was performed on the day of treatment completion and 3 months later

ELIGIBILITY:
Inclusion Criteria:

* History of BMS for at least 6 months
* no clinical changes in the oral cavity that are clinically verifiable and may affect symptoms,
* no previous BMS therapy
* age over 18

Exclusion Criteria:

* V and VII nerve neuralgia
* patients with uncontrolled diabetes mellitus,
* thyroid disease, anemia,
* Sjogren's disease and
* connective tissue disease (fibromyalgia),
* patients after prior surgical / neurosurgical treatment of the head,
* oncological treatment (radiotherapy),
* pregnant women,
* the occurrence of clinical pathologies in the oral cavity that may cause pain,
* deficiencies of vitamin B12, folic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
assessment of pain | 1 month and 3 months after therapy
  combining the use of clonazepam versus the group wearing a tongue protector Tongue protector was use in order to exclude occlusal parafunction. VAS (visual analog scale) was use to asses pain score before and after therapy
  scale from 0 to 10 0 no pain 10 maximum pain
Assessment of the depression patients diagnosed with BMS. | 1 month and 3 months after therapy
  Assessment depression Beck depresion scale Questionnaire
  scale from 0 to 28 0 no deppresion 28 depression
Assessment of the sleepiness patients diagnosed with BMS. | 1 month and 3 months after therapy
  assessment of side effects when taking clonazepam such as sleepiness was assessed on the basis of surveys with patients: Athenian Insomnia Scale Questionnaire
  scale from 0 to 24
  0 no sleep disorders 24 insomnia
assessment of side effects : slowness | 1 month and 3 months after therapy
  assessment of side effects when taking clonazepam such as dry mouth, slowness, was assessed on the basis of surveys with patients

CONTACTS AND LOCATIONS:
Overall Officials: tomasz konopka, prof, Study Director — Wroclaw Medical University
Locations (1):
- Jacek Zborowski, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No